CLINICAL TRIAL: NCT02548962
Title: A Randomized Multicenter Study of Ibrutinib in Combination With Pomalidomide and Dexamethasone in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of Ibrutinib in Combination With Pomalidomide and Dexamethasone in Subjects With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After completing Phase 1, the Sponsor elected not to move forward with Phase 2.
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCYC-1138-CA; PCI-32765 (Other: Sponsor)
Record Dates: First submitted 2015-09-03; First posted 2015-09-14 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bruton's Tyrosine Kinase; PCI-32765; Pomalidomide; Dexamethasone; Relapsed Refractory Multiple Myeloma; Ibrutinib
MeSH Terms: conditions — Multiple Myeloma | interventions — ibrutinib; pomalidomide; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase 1: Dose Finding (Experimental): Ibrutinib PO+ Pomalidomide PO+ Dexamethasone PO
  Interventions: Drug: Ibrutinib; Drug: Pomalidomide; Drug: Dexamethasone
- Phase 2: Treatment Arm A (Experimental): Ibrutinib PO+ Pomalidomide PO+ Dexamethasone PO
  Interventions: Drug: Ibrutinib; Drug: Pomalidomide; Drug: Dexamethasone
- Phase 2: Treatment Arm B (Experimental): Placebo PO+ Pomalidomide PO+ Dexamethasone PO
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Ibrutinib
  Arms: Phase 1: Dose Finding; Phase 2: Treatment Arm A
Drug: Pomalidomide
Drug: Dexamethasone
Drug: Placebo
  Arms: Phase 2: Treatment Arm B

SUMMARY:
Phase 1 is an open-label, dose finding, multicenter study of ibrutinib in combination with pomalidomide and dexamethasone in subjects with relapsed/refractory multiple myeloma.

Phase 2b is a randomized, double-blind, multicenter study of ibrutinib or placebo, in combination with pomalidomide and dexamethasone in subjects with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (Btk) is an enzyme that is present in hematopoietic cells other than T cells and is necessary for downstream signal transduction from various hematopoietic receptors including the B cell receptor as well as some Fc, chemokine, and adhesion receptors, and is crucial for both B cell development and osteoclastogenesis. Although down-regulated in normal plasma cells, Btk is highly expressed in the malignant cells from many myeloma patients and some cell lines. Ibrutinib is a potent and specific inhibitor of Btk currently in Phase 2 and 3 clinical trials. The current study is designed and intended to determine the safety and efficacy of ibrutinib in combination with pomalidomide and dexamethasone in subjects with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with relapsed/refractory MM who have received at least two prior lines of therapy including lenalidomide and either bortezomib or carfilzomib and have demonstrated disease progression on or within 60 days of the completion of the most recent treatment regimen.
* Measurable disease defined by at least ONE of the following:

  1. Serum monoclonal protein (SPEP) ≥1 g/dL.
  2. Urine monoclonal protein (UPEP) ≥200 mg by 24 hour urine.
* Adequate hematologic, hepatic, and renal function
* ECOG performance status of ≤ 2

Exclusion Criteria:

* Subject must not have primary refractory disease
* Plasma cell leukemia, primary amyloidosis or POEMS syndrome
* Unable to swallow capsules or disease significantly affecting gastrointestinal function
* Requires treatment with strong CYP3A inhibitors
* Women who are pregnant or breast feeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03; Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (5):
  - City of Hope, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- Universitätsklinikum Carl Gustav Carus, Dresden, Germany
- 'Alexandra' General Hospital of Athens, Athens, Attica, Greece
- Spain (4):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Doctor Peset, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Dose Finding (560mg): Ibrutinib PO+ Pomalidomide PO+ Dexamethasone PO
  Ibrutinib (560mg)
  Pomalidomide (4mg)
  Dexamethasone (40mg)
- Phase 1: Dose Finding (840mg): Ibrutinib PO+ Pomalidomide PO+ Dexamethasone PO
  Ibrutinib (840mg)
  Pomalidomide (4mg)
  Dexamethasone (40mg)
Period: Overall Study
Arm/Group | Phase 1: Dose Finding (560mg) | Phase 1: Dose Finding (840mg)
Started | 8 | 3
Completed | 7 | 3
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Finding (560mg) | Phase 1: Dose Finding (840mg) | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 0 | 5
  >=65 years | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 63.5 [53 to 81] | 72.7 [67 to 77] | 67.5 [53 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 2 | 8
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Greece | 3 | 0 | 3
  United States | 3 | 0 | 3
  Czechia | 2 | 2 | 4
  Australia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) According to the IMWG Response Criteria Per Investigator Assessment
Description: The overall response rate, defined as the proportion of subjects achieving a best overall response of PR or better per investigator assessment per IMWG at or prior to initiation of subsequent anticancer therapy
Time Frame: 14 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Finding (560mg) | Phase 1: Dose Finding (840mg)
Number analyzed (Participants) | 8 | 3
Participants | 3 | 1

2. Secondary Outcome: Clinical Benefit Response (CBR)
Description: The clinical benefit response, defined as the proportion of subjects achieving a best overall response of MR or better per investigator assessment per IMWG at or prior to initiation of subsequent anticancer therapy.
Time Frame: 14 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Finding (560mg) | Phase 1: Dose Finding (840mg)
Number analyzed (Participants) | 8 | 3
Participants | 4 | 2

3. Secondary Outcome: Duration of Response (DOR)
Description: The time interval between the date of initial documentation of a response and the date of first documented evidence of progressive disease, death, or date of censoring for the subjects not progressed/died. The censoring date is the last adequate tumor assessment date.
Time Frame: 14 Months
Population: Median was not reached for Phase 1: Dose Finding (560 mg). Median value provided here was the median and range (min and max).
Measure: Median (Full Range); unit: Months
Groups:
- Phase 1: Dose Finding (560 mg): Ibrutinib PO+ Pomalidomide PO+ Dexamethasone PO
  Ibrutinib (560mg)
  Pomalidomide (4mg)
  Dexamethasone (40mg)
- Phase 1: Dose Finding (840 mg): Ibrutinib PO+ Pomalidomide PO+ Dexamethasone PO
  Ibrutinib (840mg)
  Pomalidomide (4mg)
  Dexamethasone (40mg)
Arm/Group | Phase 1: Dose Finding (560 mg) | Phase 1: Dose Finding (840 mg)
Number analyzed (Participants) | 3 | 1
Months | 6.5 [5.1 to 11.8] | 7.3 [7.3 to 7.3]

ADVERSE EVENTS:
Time Frame: 14 Months
Arm/Group | Phase 1: Dose Finding (560mg) | Phase 1: Dose Finding (840mg)
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/3
Serious Adverse Events (participants affected / at risk) | 8/8 | 3/3
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Dose Finding (560mg) (N=8) | Phase 1: Dose Finding (840mg) (N=3)
Pneumonia (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Atrial Fibrilation (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardio-respiratory Arrest (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Periorbital Cellulitis (Infections and infestations) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Dose Finding (560mg) (N=8) | Phase 1: Dose Finding (840mg) (N=3)
Anaemia (Blood and lymphatic system disorders) | 6 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 0
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 0 | 1
Spontaneous Haematoma (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Mitral Valve Prolapse (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Eye Oedema (Eye disorders) | 1 | 0
Lacrimation Increased (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 5 | 2
Oedema Peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Injection Site Haemorrhage (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Peripheral Swelling (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 0
Otitis Media (Infections and infestations) | 2 | 1
Oral Herpes (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Oral Fungal Infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Steptococcal Sepsis (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 1 | 0
Radiation Skin Injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura Senile (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT02548962/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02548962/SAP_001.pdf